CLINICAL TRIAL: NCT07332910
Title: Tranexaminc Acid : Single Dose vs Placebo to Modulate Postoperative Inflammation After ACL Reconstruction : A Prospective, Randomized, Double-blind Trial
Brief Title: Study the Anti-inflammatory Effect of Tranexamic Acid When Used in Anterior Cruciate Ligament Reconstruction.
Acronym: TXA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chirec (Other)
Collaborators: Centre Hospitalier Universitaire Brugmann (Other); Erasme University Hospital (Other)
Responsible Party: Principal Investigator, matthieu clanet, Doctor, Chirec
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Chirec
Record Dates: First submitted 2025-12-17; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: ACL Reconstruction; Hemarthrosis
MeSH Terms: conditions — Hemarthrosis | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Group 1: 1 dose of tranexamic acid (15mg/kg) during induction Group 2: No tranexamic acid
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamin acid (Active Comparator): This group will receive 1 dose of tranexamic acid during the induction phase, before the surgical tourniquet
  Interventions: Drug: Tranexamic Acid (TXA)
- Placebo (Placebo Comparator): This arm will receive NaCl 0,9% at the same volume as calculated for 15mg/kg of tranexamic acid (before the surgical tourniquet)
  Interventions: Drug: Placebo (NaCl 0,9%)

INTERVENTIONS:
Drug: Tranexamic Acid (TXA) — 1 dose of Tranexamic Acid 15 mg/kg
  Other Names: TXA
  Arms: Tranexamin acid
Drug: Placebo (NaCl 0,9%) — This arm will receive NaCl 0,9% at the same volume as calculated for 15mg/kg of tranexamic acid
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Tranexamic acid (TXA) is widely used in orthopedic surgery to reduce perioperative blood loss, particularly in total hip and knee arthroplasty, due to its antifibrinolytic mechanism, low cost, broad availability, and established safety profile. Its use has recently expanded to minimally invasive procedures such as knee arthroscopy and ACL reconstruction, where postoperative hemarthrosis-rather than intraoperative bleeding-is a major cause of pain, swelling, reduced range of motion, delayed rehabilitation, and impaired early recovery.

Randomized trials and meta-analyses in arthroscopic ACL reconstruction show that TXA, administered intravenously, intra-articularly, or both, reduces postoperative hemarthrosis, joint swelling, drainage volume, and early pain, while improving early functional outcomes. These benefits are mainly short term, with no consistent long-term differences, and no increased risk of thromboembolic events. Evidence in arthroscopic meniscectomy is more limited but suggests modest improvements in early recovery, which may still be clinically meaningful given TXA's favorable risk-benefit profile.

Beyond its antifibrinolytic effects, TXA may influence inflammatory pathways by inhibiting plasmin, which is involved in complement activation and inflammatory modulation. However, existing data are conflicting, with reports of both anti- and pro-inflammatory effects depending on surgical context and dosing. Importantly, most arthroscopy studies focus on clinical outcomes rather than systemic inflammation. To date, no study has comprehensively evaluated perioperative inflammatory responses to TXA in arthroscopic knee surgery, making this low-trauma setting an ideal model to investigate its potential inflammatory effects.

DETAILED DESCRIPTION:
Over the past decade, tranexamic acid (TXA) has been widely adopted in orthopedic surgery to reduce perioperative blood loss and transfusion requirements, particularly in total hip and knee arthroplasty. TXA is a synthetic lysine analogue that inhibits the activation of plasminogen to plasmin, thereby preventing fibrin degradation and limiting fibrinolysis. Due to its low cost, wide availability, and well-established safety profile when administered intravenously, TXA is now routinely used in many countries for procedures associated with a high risk of bleeding.

In recent years, interest has expanded beyond major joint replacement toward minimally invasive orthopedic procedures, such as knee arthroscopy and anterior cruciate ligament (ACL) reconstruction. Although these procedures are generally associated with limited intraoperative blood loss, postoperative hemarthrosis remains the most frequent complication of knee arthroscopy and accounts for a substantial proportion of postoperative morbidity. Hemarthrosis has been shown to induce transient histological changes in articular cartilage and synovial tissue and is associated with increased postoperative pain, joint swelling, reduced range of motion (ROM), delayed rehabilitation, and impaired early functional recovery.

Several randomized controlled trials have investigated the role of TXA in arthroscopic knee surgery. In arthroscopic ACL reconstruction, multiple studies and subsequent systematic reviews and meta-analyses have demonstrated that TXA administration-whether intravenous, intra-articular, or combined-reduces postoperative hemarthrosis, joint swelling, drainage volume, and early postoperative pain, while improving early functional outcomes such as ROM and knee scores. These benefits appear most pronounced during the first postoperative weeks, with no consistent differences observed at longer-term follow-up. Importantly, these studies have not demonstrated an increased incidence of thromboembolic events or major complications associated with TXA use.

In the setting of arthroscopic meniscectomy, data are more limited. A double-blind randomized controlled trial evaluating intravenous TXA in routine arthroscopic meniscectomy suggested modest improvements in early functional recovery, particularly during the immediate postoperative period, despite minimal expected blood loss. Editorial commentaries and systematic reviews have emphasized that, although the absolute benefit of TXA in low-risk arthroscopic procedures may be small, even modest reductions in hemarthrosis and early inflammation may be clinically relevant given the low cost and favorable safety profile of the drug.

Beyond its antifibrinolytic properties, increasing experimental and clinical evidence suggests that TXA may exert biological effects on inflammation and coagulation pathways. Plasmin is known to play a role not only in fibrinolysis but also in the activation of the complement system and modulation of inflammatory mediators. By inhibiting plasmin generation, TXA may influence postoperative inflammatory responses. However, the available evidence remains conflicting. While some studies suggest anti-inflammatory effects, others-particularly in major orthopedic procedures such as total knee arthroplasty-have reported paradoxical increases in circulating pro-inflammatory cytokines following TXA administration.

These discordant findings highlight the complexity of the interaction between coagulation, fibrinolysis, and inflammation, and suggest that the effects of TXA on inflammatory pathways may depend on surgical context, tissue trauma, and dosing strategy. Importantly, most existing studies in arthroscopic surgery have focused primarily on clinical outcomes such as hemarthrosis, pain, and function, with very limited assessment of systemic inflammatory markers.

To date, no study has comprehensively evaluated the perioperative inflammatory response to TXA in arthroscopic knee surgery using serial cytokine measurements and integrated inflammatory burden assessment. Arthroscopic procedures, characterized by limited surgical trauma and low baseline inflammatory activation, represent an ideal clinical model to investigate the potential anti-inflammatory-or pro-inflammatory-effects of TXA in a controlled and sensitive manner.

ELIGIBILITY:
Inclusion Criteria

* Adults aged 18 years or older.
* Male or female patients scheduled for primary anterior cruciate ligament (ACL) reconstruction.
* Surgery performed under spinal anesthesia, combined with a postoperative adductor canal block for analgesia.
* American Society of Anesthesiologists (ASA) physical status I or II.
* Procedure performed by a single, standardized surgical team.
* Ability to provide written informed consent.

Exclusion Criteria

* Age under 18 years.
* Pregnancy or breastfeeding.
* Preoperative treatment with anticoagulant or antiplatelet therapy that cannot be safely discontinued.
* Known coagulation disorders or history of abnormal bleeding.
* Known hypersensitivity or allergy to tranexamic acid.
* History of seizure disorders or epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Anti-inflammatory response: Variation of IL-6 over 24 hours | 24 hours
  To evaluate the effect of a single intravenous dose of tranexamic acid on the perioperative inflammatory response, assessed by serial plasma interleukin-6 (IL-6) concentrations measured preoperatively, at 6 hours, and at 24 hours postoperatively, with quantification of the inflammatory burden using the area under the curve (AUC) over the first 24 postoperative hours.

SECONDARY OUTCOMES:
Hidden blood loss | 3 days
  To quantify hidden blood loss (HBL) using perioperative hemoglobin and hematocrit measurements obtained preoperatively, at 24 hours, and on postoperative day 3.
  Total blood loss (TBL) will be estimated using validated hematocrit-based formulas incorporating postoperative day-3 hematocrit and estimated blood volume, and hidden blood loss will be calculated as HBL = TBL - intraoperative blood loss (IBL).
Anti-inflammatory response | 24 hours
  To characterize the perioperative inflammatory profile associated with tranexamic acid administration by measuring plasma levels of TNF-α, IL-8, IFN-γ, IL-1α, IL-1β, IL-2, IL-4, IL-10, and C-reactive protein (CRP)at baseline, 6 hours, and 24 hours postoperatively.
Fibrinolysis | 24 hours
  To assess the effect of tranexamic acid on perioperative fibrinolysis, evaluated through serial measurements of D-dimer levels obtained preoperatively, at 6 hours, and at 24 hours postoperatively.
Rehabilitation score | 1 week
  - KOOS score: Knee Injury and Osteoarthritis Outcome Score - 0 (worse score) - 100 (best score).
Rehabilitation score | 1 week
  IKDC score (International Knee Documentation Committee) - evaluate impact of treatement in everyday activities: 0 (worse score) - 100 (best score).
Rehabilitation | 1 week
  Range of motion: 0-150 % (extension to flexion)
adverse effect | 1 week
  One of these described: Arterial or venous thrombosis, Seizures, Hypersensitivity reactions (including anaphylaxis), Gastrointestinal adverse effects, Acute renal failure 0 = Not described
  1 = described

CONTACTS AND LOCATIONS:
Overall Officials: Karim Touihri, Principal Investigator
Locations (1):
- Chirec Delta, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Prudovsky I, Kacer D, Zucco VV, Palmeri M, Falank C, Kramer R, Carter D, Rappold J. Tranexamic acid: Beyond antifibrinolysis. Transfusion. 2022 Aug;62 Suppl 1:S301-S312. doi: 10.1111/trf.16976. Epub 2022 Jul 14. PMID 35834488
- [Background] Alkhatib N, AlNouri M, Abdullah ASA, Ahmad Alzobi OZ, Alkaramany E, Sasaki E, Ishibashi Y. Tranexamic Acid Use in Anterior Cruciate Ligament Reconstruction Decreases Bleeding Complications: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Arthroscopy. 2022 Feb;38(2):506-518.e6. doi: 10.1016/j.arthro.2021.07.030. Epub 2021 Aug 4. PMID 34358640
- [Background] Grant AL, Letson HL, Morris JL, McEwen P, Hazratwala K, Wilkinson M, Dobson GP. Tranexamic acid is associated with selective increase in inflammatory markers following total knee arthroplasty (TKA): a pilot study. J Orthop Surg Res. 2018 Jun 18;13(1):149. doi: 10.1186/s13018-018-0855-5. PMID 29914535
- [Background] Johns WL, Walley KC, Hammoud S, Gonzalez TA, Ciccotti MG, Patel NK. Tranexamic Acid in Anterior Cruciate Ligament Reconstruction: A Systematic Review and Meta-analysis. Am J Sports Med. 2021 Dec;49(14):4030-4041. doi: 10.1177/0363546521988943. Epub 2021 Feb 25. PMID 33630652
- [Background] Fried JW, Bloom DA, Hurley ET, Baron SL, Popovic J, Campbell KA, Strauss EJ, Jazrawi LM, Alaia MJ. Tranexamic Acid Has No Effect on Postoperative Hemarthrosis or Pain Control After Anterior Cruciate Ligament Reconstruction Using Bone-Patellar Tendon-Bone Autograft: A Double-Blind, Randomized, Controlled Trial. Arthroscopy. 2021 Jun;37(6):1883-1889. doi: 10.1016/j.arthro.2021.01.037. Epub 2021 Jan 30. PMID 33529783
- [Background] Hetsroni I. Tranexamic Acid During Anterior Cruciate Ligament Reconstruction Reduced Drained Blood Volume on Day 1 and Hemarthrosis Up to Day 15 but Did Not Improve Clinical Outcomes at 3 Months. J Bone Joint Surg Am. 2019 Aug 21;101(16):1516. doi: 10.2106/JBJS.19.00514. No abstract available. PMID 31436663
- [Background] Goldstein K, Jones C, Kay J, Shin J, de Sa D. Tranexamic Acid Administration in Arthroscopic Surgery Is a Safe Adjunct to Decrease Postoperative Pain and Swelling: A Systematic Review and Meta-analysis. Arthroscopy. 2022 Apr;38(4):1366-1377.e9. doi: 10.1016/j.arthro.2021.10.001. Epub 2021 Oct 14. PMID 34655767
- [Background] Mousavi H, Akbari-Aghdam H, Entezari R. The effect of tranexamic acid injection during anterior cruciate ligament reconstruction surgery on postoperative bleeding, pain and swelling. Eur J Orthop Surg Traumatol. 2023 Apr;33(3):639-644. doi: 10.1007/s00590-022-03318-8. Epub 2022 Jul 2. PMID 35779145
- [Background] Ma R, Wu M, Li Y, Wang J, Wang W, Yang P, Wang K. The comparative efficacies of intravenous administration and intra-articular injection of tranexamic acid during anterior cruciate ligament reconstruction for reducing postoperative hemarthrosis: a prospective randomized study. BMC Musculoskelet Disord. 2021 Jan 26;22(1):114. doi: 10.1186/s12891-021-03990-7. PMID 33499848
- [Background] Felli L, Revello S, Burastero G, Gatto P, Carletti A, Formica M, Alessio-Mazzola M. Single Intravenous Administration of Tranexamic Acid in Anterior Cruciate Ligament Reconstruction to Reduce Postoperative Hemarthrosis and Increase Functional Outcomes in the Early Phase of Postoperative Rehabilitation: A Randomized Controlled Trial. Arthroscopy. 2019 Jan;35(1):149-157. doi: 10.1016/j.arthro.2018.07.050. PMID 30611343
- [Background] Cen L, Liu H, Li M, Zhang YF, Zhang HJ, Huang ZY. Intraoperative tranexamic acid reduces postoperative haemarthrosis and improves early functional outcomes in double-bundle anterior cruciate ligament reconstruction. J Orthop. 2024 Dec 10;65:51-56. doi: 10.1016/j.jor.2024.12.005. eCollection 2025 Jul. PMID 39801905
- [Background] Tan TK, Ng KT, Lim HJ, Radic R. Effect of tranexamic acid in arthroscopic anterior cruciate ligament repair: A systematic review and meta-analysis of randomised clinical trials. J Orthop Surg (Hong Kong). 2021 May-Aug;29(2):23094990211017352. doi: 10.1177/23094990211017352. PMID 34027721
- [Background] Alaia MJ, Gipsman AM. Editorial Commentary: The Benefits of Tranexamic Acid May Outweigh Risks in Arthroscopy and Sports Medicine. Arthroscopy. 2021 Apr;37(4):1334-1336. doi: 10.1016/j.arthro.2021.01.027. PMID 33812531
- [Background] Nugent M, May JH, Parker JD, Kieser DC, Douglas M, Pereira R, Lim KS, Hooper GJ. Does Tranexamic Acid Reduce Knee Swelling and Improve Early Function Following Arthroscopic Meniscectomy? A Double-Blind Randomized Controlled Trial. Orthop J Sports Med. 2019 Aug 29;7(8):2325967119866122. doi: 10.1177/2325967119866122. eCollection 2019 Aug. PMID 31497612
- [Background] Na Y, Jia Y, Shi Y, Liu W, Han C, Hua Y. Administration of Tranexamic Acid to Reduce Intra-articular Hemarthrosis in ACL Reconstruction: A Systematic Review. Orthop J Sports Med. 2022 Jan 28;10(1):23259671211061726. doi: 10.1177/23259671211061726. eCollection 2022 Jan. PMID 35111862
- [Background] Lei Y, Xie J, Huang Q, Huang W, Pei F. Additional benefits of multiple-dose tranexamic acid to anti-fibrinolysis and anti-inflammation in total knee arthroplasty: a randomized controlled trial. Arch Orthop Trauma Surg. 2020 Aug;140(8):1087-1095. doi: 10.1007/s00402-020-03442-2. Epub 2020 Apr 6. PMID 32253548